CLINICAL TRIAL: NCT00788372
Title: A Long-Term Study of JNS020QD in Patients With Chronic Pain
Brief Title: An Efficacy and Safety Study of Fentanyl in Participants With Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015583; JNS020QD-JPN-N03
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Results first posted 2013-06-26 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Fentanyl Patch
MeSH Terms: conditions — Chronic Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fentanyl (Experimental): Fentanyl transdermal patch will be applied once daily up to 4 weeks in Treatment period 1, releasing at the rate of 12.5 microgram per hour (mcg/hr), maintained for 2 days and for another 48 weeks in Treatment period 2. The dose will be increased as per Investigators' discretion in both treatment periods and the maximum applied dose will be 300 mcg/hr. Total duration of treatment is 52 weeks.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Fentanyl transdermal patch will be applied daily starting at a dose of 12.5 mcg/hr, and up to 52 weeks. Dose will be increased as per Investigator's discretion.
  Other Names: JNS020QD

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of fentanyl one-day transdermal patch (JNS020QD, patch containing a drug that is put on the skin so the drug will enter the body through the skin) in participants with chronic (lasting a long time) pain.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (conducted in more than one center) and non-comparative study of fentanyl one-day transdermal patch. The study consists of 4 periods: Screening period (3-14 days), Treatment period 1 (4 weeks), Treatment period 2 (48 weeks), Tapering period (0-6 weeks) and Follow-up period (1 week). Treatment will be initiated at 12.5 microgram per hour (mcg/hr). In both Treatment period 1 and 2, the dose will be increased as per the Investigator's discretion, ranging from 12.5 mcg/hr to 100 mcg/hr and the maximum application dose will be 300 mcg/hr. However, in Treatment period 2, the dose will be increased on 7th day before the day of medical examination (only if the participant used rescue treatment for minimum of 3 times per day for minimum of 4 days). The patch will be applied on areas including the chest, abdomen, upper arm and femoral region and replaced daily. Efficacy will primarily be evaluated by visual analog scale (VAS) score. The total duration of the study treatment will be 52 weeks. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants whose medication for chronic pain meets one of the criteria among a to e (2 or more types of opioid analgesics must not be used): a) Participants who are taking non-opioid analgesic at the normal highest dose or more for at least 14 consecutive days during 12 weeks before the informed consent, but were not continuously taking the non-opioid analgesic during 14 days before the informed consent for medical reasons such as safety b) Participants who are continuously taking an additional analgesic with a certain dosage and administration for at least 14 consecutive days before the informed consent c)Participants who are continuously taking codeine phosphate or dihydrocodeine phosphate less than 270 milligram (mg) daily (except for rescue treatment) for at least 14 consecutive days before the informed consent d) Participants who are continuously taking codeine morphine hydrochloride of oral morphine equivalent dose of less than 45 mg daily (except for rescue treatment) for at least 14 consecutive days before the informed consent (less than 30 mg daily for suppositories and less than 15 mg daily for injections) e) Participants who are continuously taking fentanyl citrate injection of less than 0.3 mg daily (except for rescue treatment) for at least 14 consecutive days before the informed consent
* Participants with chronic pain continuing for at least 12 weeks before informed consent
* Participants with an average pain intensity of greater than or equal to 50 millimeter (mm) on the Visual Analog Scale in 24-hour daily living before informed consent
* Participants who can be hospitalized to the 4th day after the initiation of patch application
* Participants who were given a sufficient explanation about the investigational product and the study and gave their own consent to participate in the study

Exclusion Criteria:

* Participants whose main cause of the pain to be assessed is considered attributable to psychogenic pain
* Participants with severe respiratory function disorders
* Participants with asthma (breathing disorder in which there is wheezing and difficulty breathing) and bradyarrhythmia (slow, irregular heartbeats)
* Participants with hepatic dysfunction function such as fulminant hepatitis (inflammation of the liver) and liver cirrhosis (serious liver disorder in which connective tissue replaces normal liver tissue, and liver failure often occurs), or renal impairment such as nephritic syndrome, acute renal failure, and chronic renal failure
* Participants with organic disorder in the brain such as brain tumor who have any of these symptoms: intracranial pressure increased, consciousness disturbance or coma and respiratory disorder

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K.,Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (23):
- Japan (23):
  - Amagasaki
  - Chūō
  - Fukuoka
  - Hiroshima
  - Izumo
  - Kanazawa
  - Kawasaki
  - Kitakyushu
  - Kobe
  - Kochi
  - Koga
  - Maebashi
  - Matsumoto
  - Minato
  - Nishinomiya
  - Ohmura
  - Ohta-Ku
  - Okayama
  - Saga
  - Sapporo
  - Shimotsuga
  - Suita
  - Ube

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 148 participants were screened, of which 142 participants entered the treatment period.
Groups:
- Fentanyl: Fentanyl transdermal patch (JNS020QD, patch containing a drug that is put on the skin so the drug will enter the body through the skin) was applied once daily up to 4 weeks in Treatment period 1, releasing at the rate of 12.5 microgram per hour (mcg/hr), maintained for 2 days and for another 48 weeks in Treatment period 2. The dose was increased as per Investigators' discretion in both treatment periods and the maximum applied dose was 300 mcg/hr. Total duration of treatment was 52 weeks.
Period: Period 1 (up to 4 Weeks)
Arm/Group | Fentanyl
Started | 142
Completed | 111
Not Completed | 31
Not completed — Adverse Event | 18
Not completed — Ineligible for transfer to period 2 | 9
Not completed — Withdrawal of informed consent | 4
Period: Period 2 (Week 4 to Week 52)
Arm/Group | Fentanyl
Started | 111
Completed | 79
Not Completed | 32
Not completed — Adverse Event | 13
Not completed — Physician Decision | 9
Not completed — Withdrawal of informed consent | 9
Not completed — Aggravated symptoms | 1

BASELINE CHARACTERISTICS:
Groups:
- Fentanyl: Fentanyl transdermal patch was applied once daily up to 4 weeks in Treatment period 1, releasing at the rate of 12.5 microgram per hour (mcg/hr), maintained for 2 days and for another 48 weeks in Treatment period 2. The dose was increased as per Investigators' discretion in both treatment periods and the maximum applied dose was 300 mcg/hr. Total duration of treatment was 52 weeks.
Arm/Group | Fentanyl
Number analyzed (Participants) | 142
Age Continuous [Mean (Standard Deviation); unit: years] | 61.4 (14.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 78

OUTCOME MEASURES:

1. Primary Outcome: Questionnaire of Opioid Withdrawal Symptoms
Description: Questionnaire of opioid withdrawal symptoms is a clinician rated 11-item scale that primarily evaluates the physical components of opioid withdrawal and is based on questions and clinical observations. The total score of questionnaire of opioid withdrawal symptoms is the sum of all individual items, with less than (<) 5 points = no withdrawal, 5 to 12 points = mild withdrawal, 13 to 24 points = moderate withdrawal, 25 to 36 points = moderately severe withdrawal and greater than (>) 36 points = severe withdrawal.
Time Frame: Week 52 or endpoint (1 week after last treatment or early discontinuation)
Population: Safety population included all the participants who received at least one patch application of the investigational product. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 140
participants
  < 5 points | 137
  >=5 to <=12 points | 2
  >=13 to <=24 points | 1
  >=25 to <=36 points | 0
  >=37 points | 0

2. Primary Outcome: Dependence Questionnaire (DQ)
Description: The DQ is a clinician rated 5-item scale that evaluates dependence on drug and based on questions (Q). Based on participant's answer to Q in questionnaire, Investigator assessed whether drug dependence occurred. It comprises 5 Q which are: continuing drug for reason other than pain, using drug in more dosage than prescribed to have effect other than treatment of pain, have ever used drug with more dosage than prescribed for other purpose, anxiety with the thought of stopping drug for reason other than aggravation of symptoms by stopping this drug and feeling to violate law to get this drug.
Time Frame: Week 52 or end point (early discontinuation)
Population: as for outcome 1
Measure: Number; unit: units on a scale
Arm/Group | Fentanyl
Number analyzed (Participants) | 140
units on a scale
  Q1:Continue to use drug for reason other than pain | 1
  Q 2: Wanted to use more dosage than prescribed | 0
  Q3: Used drug with more dosage than prescribed | 0
  Q4: Anxious with thought of stopping drug | 1
  Q5: Feeling to violate law to get this drug | 0
  Judgment by doctor: Dependent and abuse | 0
  Judgement by doctor: Not dependent and no abuse | 140

3. Primary Outcome: Pain Visual Analogue Scale Score
Description: Pain visual analog scale was used to assess the amount of pain experienced by the participant throughout the day by marking a slash through the line of a 100 millimeter (mm) scale measuring pain from "no pain (0 mm)" to "worst possible pain (100 mm)".
Time Frame: Week 52 or end point (early discontinuation)
Population: Full Analysis Set (FAS) population included all the participants with the exception of participants with violation of eligibility criteria, participants with no treatment with the patch of fentanyl and participants without efficacy data after initiation of patch application.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Fentanyl
Number analyzed (Participants) | 142
mm | 58.3 (24.72) [0 to 99]

4. Primary Outcome: Number of Participants With Pain Assessed by Categorical Scale for Pain
Description: Pain intensity was measured by assessing the average intensity of pain experienced by the participant in daily living throughout the day by 4 grades: no pain at all, mild (slightly painful, but not worried), moderate (painful, but bearable) and severe (painful and unbearable).
Time Frame: Week 52 or final evaluation (early discontinuation)
Population: The FAS population included all participants with the exception of participants with violation of eligibility criteria, participants with no treatment with the patch of fentanyl and participants without efficacy data after initiation of patch application. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 141
participants
  No pain | 1
  Mild pain | 21
  Moderate pain | 101
  Severe pain | 18

5. Primary Outcome: Number of Participants With Total Painful Time Per Day
Description: The participants assessed total painful time in 1 day by the following 5 grades: less than 4 hours, 4 hours to less than 8 hours, 8 hours to less than 12 hours, 12 hours or more and all day.
Time Frame: Week 52 or final evaluation (early discontinuation)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 141
participants
  Less than 4 hours | 17
  4 hours to less than 8 hours | 29
  8 hours to less than 12 hours | 23
  12 hours or more | 40
  All day | 32

6. Primary Outcome: Number of Participants With Quality of Sleep
Description: The quality of sleep was assessed by participants that how well they have slept from the previous assessment to current assessment time by the following 4 grades: can sleep well, can sleep moderately well, cannot sleep much and cannot sleep at all.
Time Frame: Week 52 or final evaluation (early discontinuation)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 141
participants
  Can sleep well | 28
  Can sleep moderately well | 67
  Cannot sleep much | 40
  Cannot sleep at all | 6

7. Primary Outcome: Number of Rescue Treatments
Description: Rescue treatment was used for participants with lack of analgesic efficacy, to have relief from breakthrough pain and in cases where withdrawal symptoms occur. The reference one-time rescue dose used was oral morphine 5 milligram (mg) for the investigational product fentanyl one-day transdermal patch 12.5 mcg per hr. The number of rescue treatments per day were reported.
Time Frame: Week 52 or final evaluation (early discontinuation)
Population: The FAS population included all the participants with the exception of participants with violation of eligibility criteria, participants with no treatment with the patch of fentanyl and participants without efficacy data after initiation of patch application.
Measure: Mean (Standard Deviation); unit: treatments per day
Arm/Group | Fentanyl
Number analyzed (Participants) | 142
treatments per day | 1.0 (1.13)

8. Primary Outcome: Short-Form 36-Item Health Survey (SF-36) Scores
Description: The SF-36 is 36-item form related to 8 health concepts (physical functioning, role physical, role emotional, general health, social functioning, bodily pain, vitality, mental health) and 2 summary scores (physical and mental component summary). Physical functioning, role physical and bodily pain contribute to physical component; role emotional, social functioning and mental health contribute to mental component; and social functioning, vitality, and general health contribute to both. All scores are based on a scale from 0 to 100, with higher scores defining more favorable health state.
Time Frame: Week 52 or final evaluation (early discontinuation)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fentanyl
Number analyzed (Participants) | 141
units on a scale
  Physical health (summary score) | 23.0 (17.49)
  Mental health (summary score) | 42.1 (9.82)

9. Primary Outcome: Physician's Global Assessment Scale
Description: The treating physician assessed the therapeutic efficacy of the treatment by 2 grades: effective and ineffective. Numbers of participants with effective and ineffective therapeutic efficacy with the treatment were reported.
Time Frame: Week 52 or final evaluation (early discontinuation)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 142
participants
  Effective | 106
  Ineffective | 36

10. Primary Outcome: Participants Overall Assessment
Description: The participants assessed their satisfaction with therapeutic efficacy by 5 grades: satisfied very much, satisfied, equivocal, dissatisfied and dissatisfied very much. Percentage of participants who were at least satisfied (satisfied, satisfied very much) or at least neither satisfied nor dissatisfied (dissatisfied, dissatisfied very much) were reported.
Time Frame: Week 52 or final evaluation (early discontinuation)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 141
percentage of participants
  Satisfied | 31.2 [23.7 to 39.5]
  Neither satisfied nor dissatisfied | 66.7 [58.2 to 74.4]

11. Primary Outcome: Brief Pain Inventory-Short Form (BPI-SF) Total Score
Description: The BPI-SF is a self-report questionnaire designed to assess the severity and impact of pain on daily functions. It includes pain interference score which is mean value for scores for 9 BPI-SF questions ranging between 0 (does not interfere) to 10 (completely interferes) and pain subscale score which is mean value for scores for BPI-SF questions 3 to 6 ranging between 0 (no pain) to 10 (pain as bad as can imagine). Total BPI-SF score is an average of pain interference score and pain subscale score and ranges from 0 to 10; higher score indicates more pain or pain interference.
Time Frame: Week 52 or final evaluation (early discontinuation)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fentanyl
Number analyzed (Participants) | 141
units on a scale | 5.1 (2.24)

ADVERSE EVENTS:
Time Frame: Baseline up to 7 days post last dose of study drug
Arm/Group | Fentanyl
Serious Adverse Events (participants affected / at risk) | 38/142
Other Adverse Events (participants affected / at risk) | 140/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl (N=142)
Pneumonia (Infections and infestations) | 4
Acute tonsillitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia chlamydial (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Somnolence (Nervous system disorders) | 2
Altered state of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 2
Melaena (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Sweat gland disorder (Skin and subcutaneous tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Thermal burn (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl (N=142)
Nasopharyngitis (Infections and infestations) | 35
Cystitis (Infections and infestations) | 3
Tinea pedis (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Acute tonsillitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vestibular neuronitis (Infections and infestations) | 1
Pharyngotonsillitis (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Gastroenteritis bacterial (Infections and infestations) | 1
Herpes dermatitis (Infections and infestations) | 1
Urogenital infection fungal (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Hyperprolactinaemia (Endocrine disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 18
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 10
Anxiety (Psychiatric disorders) | 4
Delirium (Psychiatric disorders) | 3
Disorientation (Psychiatric disorders) | 1
Dissociative disorder (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Somnolence (Nervous system disorders) | 78
Dizziness (Nervous system disorders) | 39
Headache (Nervous system disorders) | 12
Akathisia (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 2
Extrapyramidal disorder (Nervous system disorders) | 2
Amnesia (Nervous system disorders) | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1
Cholinergic syndrome (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Dyslalia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Parkinsonism (Nervous system disorders) | 1
Stupor (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Corneal disorder (Eye disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Motion sickness (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Bradycardia (Cardiac disorders) | 2
Atrioventricular block first degree (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 5
Flushing (Vascular disorders) | 2
Pallor (Vascular disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 73
Nausea (Gastrointestinal disorders) | 71
Vomiting (Gastrointestinal disorders) | 19
Diarrhoea (Gastrointestinal disorders) | 18
Abdominal pain upper (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 6
Toothache (Gastrointestinal disorders) | 4
Dental caries (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 3
Periodontitis (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Anorectal disorder (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1
Tongue coated (Gastrointestinal disorders) | 1
Dyschezia (Gastrointestinal disorders) | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1
Contact stomatitis (Gastrointestinal disorders) | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 18
Eczema (Skin and subcutaneous tissue disorders) | 8
Dermatitis contact (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 6
Erythema (Skin and subcutaneous tissue disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Myofascitis (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Dysuria (Renal and urinary disorders) | 10
Urinary retention (Renal and urinary disorders) | 4
Pollakiuria (Renal and urinary disorders) | 3
Bladder irritation (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Post streptococcal glomerulonephritis (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Bladder disorder (Renal and urinary disorders) | 1
Menstruation delayed (Reproductive system and breast disorders) | 1
Application site pruritus (General disorders) | 15
Pyrexia (General disorders) | 11
Thirst (General disorders) | 10
Malaise (General disorders) | 10
Feeling abnormal (General disorders) | 7
Drug withdrawal syndrome (General disorders) | 6
Oedema peripheral (General disorders) | 6
Application site erythema (General disorders) | 4
Application site dermatitis (General disorders) | 3
Chest pain (General disorders) | 3
Asthenia (General disorders) | 2
Chest discomfort (General disorders) | 2
Irritability (General disorders) | 2
Feeling cold (General disorders) | 1
Gait disturbance (General disorders) | 1
Loss of control of legs (General disorders) | 1
Oedema (General disorders) | 1
Application site urticaria (General disorders) | 1
Device failure (General disorders) | 1
Weight decreased (Investigations) | 6
Blood pressure decreased (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 3
Blood creatinine increased (Investigations) | 3
Blood urea increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 3
Liver function test abnormal (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 2
Urobilin urine present (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Monocyte count increased (Investigations) | 1
Protein total decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Electrocardiogram ST-T segment abnormal (Investigations) | 1
Protein urine present (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 6
Foot fracture (Injury, poisoning and procedural complications) | 2
Joint sprain (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 2
Thermal burn (Injury, poisoning and procedural complications) | 2
Meniscus lesion (Injury, poisoning and procedural complications) | 2
Animal bite (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 1
Heat illness (Injury, poisoning and procedural complications) | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is that the Sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the Sponsor requires.